CLINICAL TRIAL: NCT01936168
Title: Mechanochemical Endovenous Ablation (MOCA) Versus RADiofrequeNcy Ablation (RFA) in the Treatment of Primary Great Saphenous Varicose Veins: a Multicentre Randomized Trial
Brief Title: MOCA Versus RFA in the Treatment of Primary Great Saphenous Varicose Veins
Acronym: MARADONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: St. Antonius Hospital (Other); OLVG (Network); BovenIJ Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Surgeon, Rijnstate Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 839-130312
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Greater Saphenous Vein Injury
Keywords: GSV; Primary Varicose Veins; Great Saphenous Vein; Treatment
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA (Active Comparator): Radiofrequency Ablation (RFA)
  Interventions: Procedure: Radiofrequency ablation (RFA)
- MOCA (Experimental): Mechanochemical Endovenous Ablation (MOCA)
  Interventions: Device: Mechanochemical Endovenous Ablation (MOCA)

INTERVENTIONS:
Device: Mechanochemical Endovenous Ablation (MOCA) — Mechanochemical Endovenous Ablation (MOCA)for treatment of great saphenous vein incompetence
  Other Names: (MOCA)
  Arms: MOCA
Procedure: Radiofrequency ablation (RFA) — Radiofrequency ablation (RFA)for treatment of great saphenous vein incompetence
  Other Names: (RFA)
  Arms: RFA

SUMMARY:
The newly developed Mechanochemical Endovenous Ablation (MOCA) device uses a technique that combines mechanical endothelial damage using a rotating wire with the infusion of a liquid sclerosant. Heating of the vein and tumescent anesthesia are not required; only local anesthesia is utilized at the insertion site. Previously we showed that endovenous MOCA, using polidocanol, is feasible and safe in the treatment of great spahenous vein (GSV) incompetence. However, larger studies with a prolonged follow-up to prove the efficacy of this technique in terms of obliteration rates are lacking. This randomized trial was designed to compare occlusion rate, post-operative pain and complications between radiofrequency ablation (RFA: the current treatment for GSV incompetence) en MOCA.

ELIGIBILITY:
Inclusion Criteria:

* Insufficiency of the GSV
* Signed informed consent
* Patient willing to participate in follow-up scheme
* Age > 18 years
* Ultrasound criteria for endovenous treatment have been met:
* Diameter GSV between 3-12 mm
* No thrombus in the to be treated segment of the GSV

Exclusion Criteria:

* Patient not able to give informed consent
* Patient unable to present at follow-up visits
* Other treatment is more suitable
* Pregnancy and breast feeding
* Known allergy/ contra-indication for sclerotherapy
* Previous ipsilateral surgical treatment of varicose veins
* Deep venous thrombosis or lung emboli in medical history
* Anticoagulant therapy
* C5-C6 varices
* Immobilization
* Fontaine II or IV peripheral arterial disease
* Severe kidney function decline (GFS < 30 mL/min)
* Coagulation disorder or increased risk for thrombo-embolic complications(hemofilie A or B, v. Willebrand disease, Glanzmann disease, Factor VII-deficiency, idiopatic thrombocytopenic purpura, Factor V Leiden)
* Liver diseases accompanied by changes in blood coagulation, livver cirrhosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occlusion rate | up to 5 years
  Occlusion rates between treatments will be compared at mentioned time points (both technical and clinical success)

SECONDARY OUTCOMES:
Per-procedural pain score | two weeks
  Pain during the procedure will be compared between treatments using the VAS score
Complications | 30 days
  Complication at day 30 will be compared between treatments.
Procedure duration | 30 days
  The duration of the procedures will be compared
Costs of both treatments | 1 year
  The total costs of both treatments will be compared
Health status | 1 year, 5 years
  Using the RAND 36-Item short From Health Survey (SF36) the general health status will be compared between treatments at various time points as specified by the protocol.
Post procedural pain score | two weeks
  Pain during the the first two weeks after the procedure will be compared between treatments using the VAS score
Disease related quality of life | 1 year, 5 years
  Using the Aberdeen Varicose Vein Questionnaire (AVVQ)the disease related quality of life will be compared between treatments at various time points as specified by the protocol.

OTHER OUTCOMES:
Recovery time | 30 days
  Time until daily activities and or work can be resumed (measured in days)

CONTACTS AND LOCATIONS:
Overall Officials: MMPJ Reijnen, MD, Principal Investigator — Rijnstate Hospital Arnhem
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Arnhem, Gelderland
  - BovenIJ Hospital, Amsterdam
  - OLVG, Amsterdam
  - UMCG, Groningen
  - St. Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Boersma D, van Eekeren RR, Werson DA, van der Waal RI, Reijnen MM, de Vries JP. Mechanochemical endovenous ablation of small saphenous vein insufficiency using the ClariVein((R)) device: one-year results of a prospective series. Eur J Vasc Endovasc Surg. 2013 Mar;45(3):299-303. doi: 10.1016/j.ejvs.2012.12.004. Epub 2013 Jan 9. PMID 23312507
- [Background] van Eekeren RR, Boersma D, Elias S, Holewijn S, Werson DA, de Vries JP, Reijnen MM. Endovenous mechanochemical ablation of great saphenous vein incompetence using the ClariVein device: a safety study. J Endovasc Ther. 2011 Jun;18(3):328-34. doi: 10.1583/11-3394.1. PMID 21679070
- [Background] van Eekeren RR, Boersma D, Konijn V, de Vries JP, Reijnen MM. Postoperative pain and early quality of life after radiofrequency ablation and mechanochemical endovenous ablation of incompetent great saphenous veins. J Vasc Surg. 2013 Feb;57(2):445-50. doi: 10.1016/j.jvs.2012.07.049. Epub 2012 Nov 8. PMID 23141679
- [Background] van Eekeren RR, Boersma D, de Vries JP, Reijnen MM. [Endovenous mechanochemical ablation for varicose veins--a new endovenous technique without tumescent anaesthesia]. Ned Tijdschr Geneeskd. 2011;155(33):A3177. Dutch. PMID 21854655
- [Derived] Holewijn S, van Eekeren RRJP, Vahl A, de Vries JPPM, Reijnen MMPJ; MARADONA study group. Two-year results of a multicenter randomized controlled trial comparing Mechanochemical endovenous Ablation to RADiOfrequeNcy Ablation in the treatment of primary great saphenous vein incompetence (MARADONA trial). J Vasc Surg Venous Lymphat Disord. 2019 May;7(3):364-374. doi: 10.1016/j.jvsv.2018.12.014. PMID 31000063
- [Derived] van Eekeren RR, Boersma D, Holewijn S, Vahl A, de Vries JP, Zeebregts CJ, Reijnen MM. Mechanochemical endovenous Ablation versus RADiOfrequeNcy Ablation in the treatment of primary great saphenous vein incompetence (MARADONA): study protocol for a randomized controlled trial. Trials. 2014 Apr 11;15:121. doi: 10.1186/1745-6215-15-121. PMID 24726004